CLINICAL TRIAL: NCT00004663
Title: Epidemiologic Study of Reproductive Outcome in Women With Systemic Lupus Erythematosus
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Northwestern University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/11926; NU-501
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-07

CONDITIONS: Systemic Lupus Erythematosus
Keywords: arthritis & connective tissue diseases; immunologic disorders and infectious disorders; rare disease; systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis; Connective Tissue Diseases; Immune System Diseases; Communicable Diseases; Rare Diseases

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
OBJECTIVES: I. Evaluate whether pregnancy is an independent risk factor that affects disease activity in women with systemic lupus erythematosus.

II. Evaluate whether maternal disease activity is a risk factor for adverse pregnancy outcome.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a case-controlled study. Intensive data collection begins when a patient becomes pregnant.

Pregnant women are evaluated with interval pregnancy/exposure history and a clinical exam, including the Systemic Lupus Activity Measure (SLAM). Assessments are scheduled every 3 months as follows: visit 1 when the pregnancy is confirmed, visit 2 during the second trimester, visit 3 during the third trimester, visit 4 at 3 months postpartum, and visit 5 at 6 months postpartum. Visits 4 and 5 include an infant exam for growth and morphologic parameters; these visits occur on the same schedule if there is a miscarriage or stillbirth.

Patients not currently pregnant are randomly chosen to be followed as controls. These patients undergo a review of current pregnancy status and measures of disease activity, including SLAM, every 3 months for 5 visits.

ELIGIBILITY:
* Definite or probable systemic lupus erythematosus meeting American College of Rheumatology criteria

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 480
Dates: Start 1994-02

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind Ramsey-Goldman, Study Chair — Northwestern University